CLINICAL TRIAL: NCT01830218
Title: A National Survey on Obstetric Anesthesia and Analgesia Care in Czech Republic
Brief Title: Obstetric Anesthesia and Analgesia Month Attributes in Czech Republic
Acronym: OBAAMA
Status: Completed | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Collaborators: Masaryk University (Other); General University Hospital, Prague (Other); Brno University Hospital (Other)
Responsible Party: Principal Investigator, Jan Blaha, MD, PhD., Chairman, ESPAA, Charles University, Czech Republic
Other Study IDs: OBAAMA 2011
Record Dates: First submitted 2013-04-07; First posted 2013-04-12 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2013-04

CONDITIONS: Obstetric Anesthesia Care
MeSH Terms: interventions — Anesthesia, Obstetrical; Analgesia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Obstetric anesthesia and analgesia: Women in labor undergoing anesthesia care
  Interventions: Procedure: Obstetric anesthesia and analgesia

INTERVENTIONS:
Procedure: Obstetric anesthesia and analgesia — All anesthesia procedures during labor: labor analgesia, anesthesia for Cesarean section, anesthesia for procedures in third stage of labor

SUMMARY:
A national survey of current practices, preferred drug and technique choices for obstetric anesthesia and analgesia in Czech Republic.

DETAILED DESCRIPTION:
A one month-long project monitoring an obstetric anesthesia practices in obstetric/anesthesia departments throughout the Czech Republic.

Electronic Case Report Form (eCRF) is used to collect data on all obstetric anesthesia procedures in peripartal period and obstetric and anesthesia complications. All consecutive cases in each participating center during the study period are recorded. Each record is related to parturient and contains the following sections: history, form of labour analgesia, type of anesthesia for Cesarean section and anesthesia in third stage of labor.

ELIGIBILITY:
Inclusion Criteria:

Women in labor undergoing anesthesia care

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women in labor
Sampling Method: Non-Probability Sample
Enrollment: 1940 (Actual)
Dates: Start 2011-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
A national survey of current practice of obstetric anesthesia and analgesia in Czech Republic | Parturition period, up to 24 hours after labor
  Monitoring of all obstetric anesthesia procedures in peripartal period and anesthesia complications: history, form of labour analgesia, type of anesthesia for Cesarean section and anesthesia in third stage of labor.

CONTACTS AND LOCATIONS:
Overall Officials: Petr Stourac, MD, PhD., Study Chair — ESPAA
Locations (1):
- University Hospital Brno, Brno, Czechia

REFERENCES:
- See also: Study webpage — http://obaama.registry.cz/